CLINICAL TRIAL: NCT00818844
Title: Role of Nepafenac in Reducing Macular Volume After Epiretinal Membrane Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SMA-08-10
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2012-02

CONDITIONS: Epiretinal Membrane
Keywords: Nepafenac; vitrectomy surgery; Epiretinal membrane surgery
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nepafenac (Experimental): Nepafenac 0.1% dosed topically TID for 3 months after Epiretinal Membrane (ERM) Surgery
  Interventions: Drug: Nepafenac 0.1%
- BSS (Placebo Comparator): BSS dosed topically TID for 3 months after Epiretinal Membrane (ERM) Surgery
  Interventions: Other: BSS

INTERVENTIONS:
Drug: Nepafenac 0.1% — NSAID
  Arms: Nepafenac
Other: BSS — BSS
  Arms: BSS

SUMMARY:
The purpose of this study is to compare the macular volume of patients treated with a 3-month course of topical Nepafenac (0.1% solution) to patients treated with a placebo course following epiretinal membrane surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 year of age or older, of any race and either sex.
* Able to understand and sign an informed consent that has been approved by an Institutional Review Board.
* Must agree to comply with study visit schedule and other study requirements.
* Must have vision loss associated with idiopathic epiretinal membrane and secondary retinal edema.
* Must have pre-operative central foveal thickness greater than 300 microns.
* Prior cataract surgery must be at least 6 months postoperative.

  * Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Vision loss associated with maculopathies other than idiopathic epiretinal membrane and secondary retinal edema (e.g. branch retinal vein occlusion, central retinal vein occlusion, wet macular degeneration, diabetic retinopathy, posterior uveitis).
* Dry macular degeneration (drusen) with central geographic atrophy.
* Concomitant cataract surgery performed at the time of study vitrectomy.
* Prior vitrectomy surgery in the study eye(s).
* Prior macula laser treatment in the study eye(s).
* Prior periocular steroid injections in the study eye(s) within preceding 6 months.
* Prior cataract surgery in the study eye(s) within the last 6 months.
* Any systemic or ocular disease or disorder, complicating factors or structural abnormality that would negatively affect the conduct or outcome of the study.
* Use of topical ocular medications during the study period.
* Antibiotics (systemic or topical) outside of study protocol may not be used within 7 days of preoperative/baseline visit or anytime after this visit for the duration of the study.
* Women of childbearing potential not using reliable means of birth control.
* Women who are pregnant or lactating.
* Enrollment of more than one person per household at the same time.
* Enrollment of the investigator or his or her staff, family members of the investigator, family members of the investigator's staff, or individuals living in the households of these individuals.
* Participation in any investigational drug or device study within 30 days of entering this study. Note: Patients may have both eyes enrolled in this study provided that 2nd eye enrollment takes place 30 days after completion of the first eye. Second eye will receive the same study treatment as first eye.

  * Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Macular thickness | 12 weeks post operative
  Macular thickness as measured by SD-OCT

SECONDARY OUTCOMES:
Visual Acuity | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dan Miller, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Schoenberger SD, Miller DM, Petersen MR, Foster RE, Riemann CD, Sisk RA. Nepafenac for epiretinal membrane surgery. Ophthalmology. 2011 Jul;118(7):1482.e1-3. doi: 10.1016/j.ophtha.2011.01.034. No abstract available. PMID 21724047